CLINICAL TRIAL: NCT01811108
Title: Assessment of Clinical Practice Administration of Chemotherapy and Anti-angiogenic Agent (Bevacizumab) Retrospectively (From 1/7/2009) and Prospectively (up to 31/12/2013) as First Line Treatment for Patients With Locally Advanced or Metastatic Colorectal Cancer (With or Without KRAS Mutation). Assessment of Toxicity, Compliance and Survival of Patients.
Brief Title: Assessment of Clinical Practice Administration of Chemotherapy and Anti-angiogenic Agent (Bevacizumab) in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: CT/10.12
Record Dates: First submitted 2013-02-21; First posted 2013-03-14 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: mCRC; KRAS mutation; Chemotherapy; Anti-angiogenic agent; Bevacizumab; 1st Line
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Avastin regimens: Patients who have either received or who are going to receive chemotherapy plus Avastin (bevacizumab)

SUMMARY:
Investigators propose to assess, retrospectively (from 1/7/2009) and prospectively (up to 31/12/2013,) the safety and tolerability profile (number of participants with adverse events) of standard chemotherapy and anti-angiogenic agent bevacizumab (Avastin) as first line treatment of patients with metastatic Colorectal Cancer with or without KRAS mutation. All treatment schedules that are going to be assessed are considered by the international guidelines as standard therapy for patients with metastatic Colorectal Cancer.

DETAILED DESCRIPTION:
In addition investigators propose to assess the compliance of patients to treatment and the efficacy of treatment. That means percentage of objective responses, duration of response, frequency of curative liver resection after the administration of treatment, progression free survival and estimation of overall survival

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically confirmed metastatic or locally advanced non-operable colorectal cancer
* No prior first line treatment for metastatic colorectal cancer
* Age ≥18 years
* One or more measurable lesions (≥1cm in diameter with spiral CT scan or ≥2cm with conventional techniques) according to RECIST criteria
* ECOG performance status ≤2
* Adequate haematological, renal and hepatic function
* Urine protein <2+ (dipstick)
* Life expectancy of ≥12 weeks

Exclusion Criteria:

* Previous first line treatment for metastatic colorectal cancer(progression >6 months after the end of adjuvant treatment)
* Previous radiotherapy to target lesions
* Patients with brain metastases and/or cancerous meningitis
* Metastatic infiltration >50% of the liver parenchyma
* Presence or history of other neoplasm except properly treated basal cell skin cancer or in situ cervical carcinoma
* Patients participating in interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinics for cancer prevention
Sampling Method: Probability Sample
Enrollment: 670 (Actual)
Dates: Start 2009-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with AE | Every 2 weeks up to 12 weeks
  In this observational study investigators are going to assess standard schedules in which administration was every 2 weeks.

SECONDARY OUTCOMES:
Number of Participants with Response Rate | Disease evaluation at Week 6
  In this observational study investigators are going to assess standard schedules in which the disease evaluation was performed every 6 weeks
Percentage of Patients with Progression Free Survival | 1 year
Patients Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — Hellenic Oncology Research Group
Locations (6):
- Greece (6):
  - University Hospital of Crete, Dep of Medical Oncology, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dept. of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki